CLINICAL TRIAL: NCT00486941
Title: A Randomized Trial of Lifestyle Intervention in Primary Health Care for the Modification of Cardiovascular Risk Factors - the Björknäs Study
Brief Title: Lifestyle Intervention in Primary Health Care - the Björknäs Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: County Council of Norrbotten, Sweden (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPN-Umea 02-512
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Hypertension; Type 2 Diabetes; Obesity; Dyslipidemia
Keywords: Primary Prevention; Health Promotion; Diet; Exercise; Risk Factors; Randomized Controlled Trial
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Obesity; Dyslipidemias; Motor Activity | interventions — Exercise; dentin sialophosphoprotein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Exercise and diet - based on DPS and DPP

SUMMARY:
The purpose of this study is to determine whether a short group intervention programe aiming at lifestyle changes at a local health centre can improve risk factors for cardiovascular disease

DETAILED DESCRIPTION:
Successfully transferring the findings of expensive and tightly controlled lifestyle intervention programmes to the primary care setting is necessary if such knowledge is to be used for disease prevention at the population level. Therefore, our objective was to evaluate the efficacy of a lifestyle intervention programe in the primary health care setting, targeted at patients with moderate- to high-risk of cardiovascular disease according to cardiovascular risk factor levels, physical activity and quality of life ratings.

Randomised controlled trial with follow-up at 3, 12, 24 and 36 months, carried out in a primary health care centre in Northern Sweden. A total of 151 middle-aged men and women, with hypertension, dyslipidemia, type 2 diabetes or obesity were enrolled. The subjects were randomised to an intervention (n = 75) or control group (n = 76). 120 subjects completed the three-year follow-up. The intervention was based on the protocols used in the Finnish Diabetes Prevention study (DPS) and the U.S Diabetes Prevention Program

ELIGIBILITY:
Inclusion Criteria:

* Patients from one single health care centre with a diagnosis of:

  * Typ 2 diabetes,
  * Hypertension,
  * Obesity or
  * Dyslipidemia

Exclusion Criteria:

* Coronary heart
* Disease,
* Stroke,
* TIA,
* BP >180/105,
* Dementia; or
* Severe psychiatric disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2003-02; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Changes in anthropometry (BMI, waist and hip cf) | 3 years
Maximal oxygen uptake (VO2max) | 3 years
Health-related quality of life (EQ 5D, SF-36) | 3 years
Self-reported physical activity | 3 years

SECONDARY OUTCOMES:
Blood pressure | 3 years
Total cholesterol, HDL and triglycerides | 3 years
Glucose tolerance (OGTT) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mats CE Eliasson, MD, PhD, Principal Investigator — Umeå University, Umeå, Sweden
Locations (1):
- Björknäs Health Centre, Boden, Sweden

REFERENCES:
- [Result] Eriksson KM, Westborg CJ, Eliasson MC. A randomized trial of lifestyle intervention in primary healthcare for the modification of cardiovascular risk factors. Scand J Public Health. 2006;34(5):453-61. doi: 10.1080/14034940500489826. PMID 16990155
- [Derived] Eriksson MK, Hagberg L, Lindholm L, Malmgren-Olsson EB, Osterlind J, Eliasson M. Quality of life and cost-effectiveness of a 3-year trial of lifestyle intervention in primary health care. Arch Intern Med. 2010 Sep 13;170(16):1470-9. doi: 10.1001/archinternmed.2010.301. PMID 20837834
- [Derived] Eriksson MK, Franks PW, Eliasson M. A 3-year randomized trial of lifestyle intervention for cardiovascular risk reduction in the primary care setting: the Swedish Bjorknas study. PLoS One. 2009;4(4):e5195. doi: 10.1371/journal.pone.0005195. Epub 2009 Apr 14. PMID 19365563